CLINICAL TRIAL: NCT06654245
Title: Toward an Integrated Approach to Assessing and Addressing Follow-Up Care Needs That Will Facilitate Care Transitions for Cancer Survivors: A Pilot Study
Brief Title: Assessing and Addressing Follow-up Care Needs That Will Facilitate Care Transitions for Cancer Survivors
Acronym: SHAREDCare
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accruals, PI decision
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00119287; P30CA012197 (NIH); ONC-LUN-2403 (Other: AHWFBCCC)
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Stage I Lung Cancer; Stage II Lung Cancer; Stage III Lung Cancer; Stage IV Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHAREDCare Supportive care arm (Experimental): Patients receive a SHAREDCare call with a navigator to discuss identified distress and social needs and develop/deploy a shared response plan to address identified needs on study. Patients also receive standard of care automated referrals on study. Two weeks following the initial call, patients receive a second SHAREDCare call with a navigator to follow-up on the shared response plan.
  Interventions: Behavioral: Telephone based interview; Other: Survey using a questionnaire.; Other: Electronic health record review; Other: Referral

INTERVENTIONS:
Behavioral: Telephone based interview — Receive SHAREDCare navigator calls
Other: Survey using a questionnaire. — Ancillary studies
Other: Electronic health record review — Ancillary studies
Other: Referral — Receive standard of care automated referrals

SUMMARY:
This clinical trial evaluates whether a shared response plan (SHAREDCare) improves follow-up care for lung cancer survivors. As the number of cancer survivors increases, there is a new need for high-quality chronic illness care. High-quality chronic illness care can be difficult to deliver and involves working with the patient to be certain they have what they need to be actively involved with their care to meet their needs. SHAREDCare allows the patient to work with a navigator to review identified distress and social needs. The patient and navigator discuss the needs and develop a shared response plan to address the needs in ways that consider the patient's current behaviors, beliefs, and motivation. The plan also establishes specific patient goals, anticipates barriers, and establishes how the navigator will follow-up on the needs and adjust care and assistance when needed. Using a shared response plan may improve follow-up care for lung cancer survivors.

DETAILED DESCRIPTION:
Primary Objective: Pilot and qualitatively assess the acceptability of SHAREDCare through semi- structured interviews

Secondary Objectives:

* Describe quantitative assessments of intervention acceptability, appropriateness, and feasibility.
* Describe survivor level of unmet needs13 using a validated measure to collect data before and/or after completion of the SHAREDCare intervention.
* Track clinical referrals and other actions made as a result of patient responses on the Electronic Distress Screening (EDS) and the percentage of referrals that have been "completed" (i.e. those referrals where a patient completed the relevant medical or social needs-related visit).
* Track recruitment, assessment completion, and any related adverse events.

OUTLINE:

Patients receive a SHAREDCare call with a navigator to discuss identified distress and social needs and develop/deploy a shared response plan to address identified needs on study. Patients also receive standard of care automated referrals on study. Two weeks following the initial call, patients receive a second SHAREDCare call with a navigator to follow-up on the shared response plan.

After completion of study intervention, patients are followed up 4 weeks after initial call.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed study disease. A pathology report should be referenced/available (stages I-IV lung cancer)
* Ability to understand and the willingness to sign an institutional review board (IRB)-approved informed consent document
* ≥ 18 years of age
* Within two years of lung cancer diagnosis
* Able to understand, read and write English

Exclusion Criteria: Does not meet the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-01-12 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
SHAREDCare's Qualitative Acceptability | At 4 weeks post-initial call
  Will be assessed with semi-structured interviews. These methods will be guided by Grounded Theory, a process using inductive coding to develop theory from data (e.g., themes relating to components, timing, or delivery of the intervention).

SECONDARY OUTCOMES:
SHAREDCare's Quantitative Acceptability | At 4 weeks post-initial call
  Will be measured with the Acceptability of Intervention Measure. Quantitative analyses will include descriptive statistics of quantitative data on level of clinical and demographic characteristics and acceptability. Distributions of continuous variables (acceptability) will be examined for estimation of standard deviations (SD) that will be used to inform power analysis for future studies.
SHAREDCare's Quantitative Appropriateness | At 4 weeks post-initial call
  Will be measured with the Intervention Appropriateness Measure. Quantitative analyses will include descriptive statistics of quantitative data on level of clinical and demographic characteristics and appropriateness. Distributions of continuous variables (acceptability) will be examined for estimation of SD that will be used to inform power analysis for future studies.
SHAREDCare's Quantitative Feasibility | At 4 weeks post-initial call
  Will be measured with the Feasibility Intervention Measure. Quantitative analyses will include descriptive statistics of quantitative data on level of clinical and demographic characteristics and feasibility. Distributions of continuous variables (acceptability) will be examined for estimation of SD that will be used to inform power analysis for future studies
Number of Survivors With Unmet Needs | At baseline and at 4 weeks post-initial call
  Will be assessed before and/or after completion of the SHAREDCare intervention using a validated measure called the Survivor Unmet Needs Survey. This measure will be used to determine the prevalence and predictors of cancer survivors' unmet needs. Scores at baseline and follow-up will be summarized as median (interquartile range, range). Changes will be tested by Wilcoxon signed-rank test.
Number of Clinical Referrals Made | At 4 weeks post-initial call
  Quantitative analyses will include descriptive statistics of quantitative data on level of clinical and demographic characteristics and referrals.
Percentage of Referrals Completed | At 4 weeks post-initial call
  Will be defined as those referrals where a patient self-reported completing the relevant visit documented in a format adapted from another study. Quantitative analyses will include descriptive statistics of quantitative data on level of clinical and demographic characteristics and referrals.
Number of Participants Enrolled/Eligible | At 4 weeks post-initial call
  The number of eligible participants will be tracked and for those not enrolled, reasons will be summarized. Will calculate the percent of participants who complete the follow-up visit to assess retention. Will also compare demographic characteristics and baseline scores of participants who complete the follow-up visit to those who do not via Fisher's exact tests or Wilcoxon rank sum tests as appropriate.
Percentage of Assessments Completed | At 4 weeks post-initial call
  The percent of participants who complete the follow-up visit to assess retention. Will also compare demographic characteristics and baseline scores of participants who complete the follow-up visit to those who do not via Fisher's exact tests or Wilcoxon rank sum tests as appropriate.
Number of Adverse Events Reported | At baseline (initial call) up to 4 weeks post-initial call
  The frequency of any adverse events will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Atrium Health Wake Forest Baptist Comprehensive Cancer Center (AH-WFBCCC), Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-07-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT06654245/ICF_000.pdf